CLINICAL TRIAL: NCT05174546
Title: Performance of Emerging Microbiological Techniques for the Diagnosis of Severe Infections in Neutropenic Patients With Haematological Malignancies
Brief Title: New Diagnostics in Neutropenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Other Study IDs: HREC/2021/QRBW/78988
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Febrile Neutropenia
MeSH Terms: conditions — Febrile Neutropenia | interventions — Magnetic Resonance Myelography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: T2 magnetic resonance — Samples for assessment by the T2MR will be collected once daily in occasion of any consecutive febrile episode during neutropenia when blood cultures are ordered as per standard of care. T2 magnetic resonance will be run according to manufacturer's instructions

SUMMARY:
Mortality due to bloodstream infections in patients with neutropenia and haematological malignancies is high and optimal management is hampered by long turnaround times of conventional blood cultures.

This is an observational study to assess the performance of T2 magnetic resonance, in diagnosing proven, probable and possible bloodstream infections as well as its theoretical impact on antimicrobial prescriptions in neutropenic patients with acute leukemia and bone marrow recipients.

DETAILED DESCRIPTION:
Study Background

In patients with haematological malignancies, neutropenia often leads to the development of severe infections, including bloodstream, which are characterized by high mortality. Patients' management can be challenging as conventional diagnostic methods for the diagnosis of such infections are affected by several limitations, including limited sensitivity and long turnaround time.

T2 Magnetic Resonance (T2MR) is a new technology able to identify pathogens directly from whole blood in few hours, and preliminary data showed how it might have higher sensitivity compared to blood cultures.

Study Aims

* To assess the performance of the T2MR (including the T2Candida, T2Bacteria and T2Resistance) in diagnosing proven, probable, and possible bloodstream infection (BSI) due to T2 on-panel pathogens, in patients affected by haematological malignancies with febrile neutropenia, including patients with acute leukaemia and bone marrow transplant recipients.
* To assess the mean time to results of the T2MR 3 panels as compared to blood cultures. These will be considered as an estimate of time to optimal treatment in proven, probable, and possible BSI.
* To estimate the potential impact of T2MR results on antimicrobial modifications in neutropenic patients with proven/probable and possible BSI.

Methods

Prospective observational study. Patients with acute leukemia or bone marrow transplant recipients and febrile neutropenia, admitted to the Haematology ward, will be consecutively enrolled in the study. 100 consecutive febrile episodes will be included in the study.

At the time of blood culture collection (ordered as per standard of care), blood samples for T2MR (including T2Bacteria, T2Candida and T2Resistance) will be also collected.

The performance of the T2 assays will be compared to that of proven, probable, and possible BSI defined by standard of care laboratory practices due to T2 on-panel pathogens, and time to results will be assessed as an estimate of time to optimal treatment.

Moreover the potential impact of T2 positive results on antimicrobial modifications will be estimated including escalation, de-escalation and antimicrobial change.

Proven BSI is defined by a positive blood culture; probable BSI is defined by a negative blood culture but a positive T2 result if the T2-detected organism is isolated within 21 days from another clinical specimen; possible BSI is defined as a negative blood culture but a positive T2 result in the absence of supporting culture data if the T2-detected organism or resistance gene was a plausible cause of infection.

Data analysis

Sensitivity, specificity, and predictive values will be calculated using proven, probable, and possible BSI as a reference, with 95% confidence intervals.

Mean time to T2 results will be compared to mean time to blood cultures results.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (> 18 years old) affected by acute leukaemia and/or recipients of bone marrow transplantation for any disease indication (during the pre and post-transplant phase) who develop febrile neutropenia, where blood cultures (and possibly bronchoscopy) are ordered as per standard of care.

Febrile neutropenia is defined as:

* an ANC of <500 cells/mm3
* a single temperature measurement of ≥38.0°C

Exclusion Criteria:

* Patients not able to provide informed consent
* Death is deemed imminent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by acute leukemia and bone marrow transplant recipients who are admitted to the Haematology Unit and are expected to encounter chemotherapy-induced or pre/post-transplant neutropenia during the course of hospital admission, will be approached by research staff to discuss participation. Study aims and design will be discussed and the opportunity to read the Patient Information and Consent Form and ask questions will be provided. Patients or their representative will be provided an informed consent form to confirm participation, and consent will be obtained prior to episodes of febrile neutropenia.
  In consenting patients, in the subsequent case of febrile episodes during neutropenia, the collection of blood samples for T2MR assessment will be performed in addition to blood cultures ordered as per standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of T2MR as compared to Blood Cultures for the diagnosis of proven, probable, and possible BSI as previously defined | 01/04/2022 - 31/03/2023
  Sensitivity and specificity of T2 magnetic resonance will be calculated with 95% confidence intervals both for pathogen identification and resistance markers detection

SECONDARY OUTCOMES:
In patients with positive T2 results: Mean time to result of T2MR | 01/04/2022 - 31/03/2023
  In patients with positive T2 results, the theoretical mean time to T2 results (if T2 assessment had been performed real time as part of the clinical laboratory workflow) will be assessed.
In patients with positive T2 results: percentage of potential antimicrobial modifications according to T2 results | 01/04/2022 - 31/03/2023
  In the case of positive T2 results, the impact of T2 results on potential antimicrobial treatment modification will be assessed. Specifically, the percentage of cases where an early T2 result would be useful for antimicrobial modification out of all the febrile episodes will be evaluated. Antimicrobial treatment changes considered will be:
  * De-escalation of treatment (replacing current treatment with an antimicrobial with narrower spectrum)
  * Escalation of treatment (replacing current treatment with an antimicrobial with broader spectrum)
  * Change of antimicrobials (replacing current treatment with an antimicrobial with similar spectrum, i.e. from vancomycin to daptomycin in case of detection of van gene)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brisbane Hospital, Brisbane, Queensland, Australia